CLINICAL TRIAL: NCT03411148
Title: Targeting Balance Confidence as a Strategy to Increase Integration and Improve Outcomes in Users of Lower-Limb Prostheses
Brief Title: Targeting Balance Confidence to Increase Community Integration in Users of Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Northwestern University (Other); Captain James A. Lovell Federal Health Care Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Noah Rosenblatt, Assistant Professor, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP160044; W81XWH-17-1-0697 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-01-10; First posted 2018-01-26 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Amputation; Physical Activity
Keywords: fear avoidance; cognitive behavioral therapy; physical therapy; prosthetic; fear of falling; gait
MeSH Terms: conditions — Motor Activity | interventions — Physical Therapists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group A (Experimental): Weekly exercise sessions with physical therapist and psychologist
  Interventions: Behavioral: Weekly exercise sessions with physical therapist and psychologist
- Exercise Group B (Placebo Comparator): Home-based exercises
  Interventions: Behavioral: Home-based exercises

INTERVENTIONS:
Behavioral: Weekly exercise sessions with physical therapist and psychologist — Eight weekly sessions integrating techniques from physical therapy and cognitive behavioral therapy. At the start of each session participants play virtual reality games that target balance and functional gait and then discuss their balance confidence and activity avoidance behaviors with a behavioural counselor. Weekly homework assignments ask participants to report on thoughts causing them to avoid activities and to slowly engage in activities that present increasing levels of fear.
  Arms: Exercise Group A
Behavioral: Home-based exercises — Stretching and other exercises are safely taught by physical therapist and then practiced at home following a provided schedule. Participants receive periodic calls to discuss progress.
  Arms: Exercise Group B

SUMMARY:
Low balance confidence occurs when an individual perceives they have limited ability to maintain their balance while performing a specific task of daily living. It is a prevalent problem in lower limb prosthesis users and is a strong predictor of prosthesis use and community participation. Balance confidence is not necessarily related to functional abilities. It is possible to improve functional ability as a result of rehabilitation, without concurrently improving balance confidence. Interventions to address low balance confidence may need to target both functional abilities as well as beliefs regarding these abilities. The purpose of this study is to test whether, for users of lower limb prostheses, an intervention combining physical therapy exercise to improve function with cognitive behavioral therapy to address fears and thoughts associated with low confidence can improve balance confidence and promote community participation.

DETAILED DESCRIPTION:
Lower limb prosthesis users, with self-reported low balance confidence complete baseline gait analysis and balance testing, as well as a series of validated self-reported outcome scales addressing balance confidence, quality of life, and community integration. Participants are then provided a step activity monitor (SAM) and a global position sensing (GPS) tracker to be worn for one week, the data from which is linked and used to objectively quantify baseline community participation. At the conclusion of the one week, participants are randomized to one of two groups, each of which will last for 8 weeks. At the conclusion of the eight weeks, participants repeat baseline assessments and are again provided a SAM and GPS tracker to wear for one week. Baseline measures and activity monitoring occur again 8 and 16 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* unilateral lower limb amputation without serious complications
* at least 6 months experience using a definitive lower limb prosthesis
* Activity Specific Balance Confidence (ABC) scale score≤80
* self-reported concern about balance that limit activities

Exclusion Criteria:

* active wounds on weight bearing surfaces
* inability to perform the protocol without an assistive device
* currently seeing a physical therapist for any reason
* history of neurodegenerative disease
* history of stroke
* ill-fitting or ill-functioning prosthesis (to be verified by research prosthetist during screening)
* prohibited by primary care physician or research physician to participate in mild exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Community integration | 24 weeks
  number of steps taken outside of the home

SECONDARY OUTCOMES:
Social Functioning scale from the 36-item Short Form Health Survey | 24 weeks
  The scale measures the extent to which physical and emotional problems interfere with social activities on a scale of 0-100 with higher scores indicating less interference
Role Limitation due to Emotional Problems scale from the Short Form Health Survey (SF36) | 24 weeks
  The scale measures the extent to which emotional problems interfere with work and daily activities on a scale of 0-100 with higher scores indicating less interference
Extent of Participation scale from the Measure of Community Reintegration of Servicemembers | 24 weeks
  The scale measures community participation in terms of how often an individual engages in certain activities on a score of 10-70 with higher scores indicating greater participation
Perceived Limitation scale from the Measure of Community Reintegration of Servicemembers | 24 weeks
  The scale measures self-perceived limitations in community participation n a score of 10-70 with higher scores indicating less limitation
Frenchay Activity Index | 24 weeks
  This is a behavioral scale that primarily measures social participation, as well as daily activities on a score of 0-45 with higher scores indicating greater social activity.
Change from baseline in Activity-specific balance confidence scale following the intervention | 8 weeks
  The ABC scale measures balance confidence on a scale of 0-100 with higher values indicating greater confidence
Activity-specific balance confidence scale | 24 weeks
  The ABC scale measures balance confidence on a scale of 0-100 with higher values indicating greater confidence. Measurement at this time point will indicate the lasting impact of the intervention on balance confidence

OTHER OUTCOMES:
Well-being scale from the Prosthetic Evaluation Questionnaire | 24 weeks
  The scale measures overall quality of life on a score of 0-100 with higher scores indicating increased quality of life.
Change from baseline in Berg Balance Scale | 8 wks
  This scale measures measures balance function by assessing the performance of functional tasks. It is scored from 0-45 with high scores indicating better balance.
Change from baseline on L-test performance | 8 wks
  Participants rise from a chair without armrests, walk 3m, turn right, walk 7m, turn around and trace their path back to the start. Time to complete the task is noted.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Rosalind Franklin University of Medicine and Science, North Chicago, Illinois

REFERENCES:
- [Derived] Rosenblatt NJ, Schneider KL, Miller SA, Hagopian K, Hagg S, Reddin C, Churchill R, Dams GM, Calamari JE, Stachowiak A, Major MJ. Mixed methods analysis of an interdisciplinary intervention to promote balance confidence in lower limb prosthesis users. Front Rehabil Sci. 2025 Sep 1;6:1626051. doi: 10.3389/fresc.2025.1626051. eCollection 2025. PMID 40959746
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273
- [Derived] Bourque MO, Schneider KL, Calamari JE, Reddin C, Stachowiak A, Major MJ, Duncan C, Muthukrishnan R, Rosenblatt NJ. Combining physical therapy and cognitive behavioral therapy techniques to improve balance confidence and community participation in people with unilateral transtibial amputation who use lower limb prostheses: a study protocol for a randomized sham-control clinical trial. Trials. 2019 Dec 30;20(1):812. doi: 10.1186/s13063-019-3929-8. PMID 31888708